CLINICAL TRIAL: NCT04869228
Title: A Phase 3 Randomized, Double-Blind Placebo Controlled, Multi-regional Trial to Evaluate the Efficacy and Safety of GT0918 for the Treatment of Mild to Moderate COVID-19 Male Patients
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: This decision is made on changing the development strategy of GT0918 to adapt ever-changing COVID-19 pandemic management globally.
Sponsor: Suzhou Kintor Pharmaceutical Inc, (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GT0918-MR-3001
Record Dates: First submitted 2021-04-29; First posted 2021-05-03 (Actual); Last update posted 2023-08-18 (Actual); Status verified 2023-08

CONDITIONS: COVID-19
Keywords: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — proxalutamide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- GT0918 in the treatment arm (Experimental): GT0918 tablets : oral, 1 time / day, 2 tablets / time, after meals
  Interventions: Drug: GT0918 tablets or placebo
- Placebo in the placebo arm (Placebo Comparator): placebo : oral, 1 time / day, 2 tablets / time, after meals
  Interventions: Drug: GT0918 tablets or placebo

INTERVENTIONS:
Drug: GT0918 tablets or placebo — GT0918 tablets or placebo: oral, 1 time / day, 2 tablets / time, after meals

SUMMARY:
The purpose of this study is to assess the efficacy and safety of Proxalutamide (GT0918) in male outpatients with mild to moderate COVID-19 disease

DETAILED DESCRIPTION:
The subjects in the experimental group will receive GT0918 (200mg oral once-daily (QD) for 14 consecutive days) in addition to supportive treatment. The subjects in the control group will receive placebo (200mg oral once-daily (QD) for 14 consecutive days) in addition to supportive treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Adult males age ≥18 years of age at the time of randomization
2. Are currently not hospitalized for acute respiratory symptoms (not applicable for subjects whose countries require mild to moderate COVID-19 patients to be hospitalised, such as COVID-19 patients in mainland China)
3. The subject's first positive SARS-CoV-2 viral infection test result (using an approved molecular test, or other approved commercial or public health assay on any approved specimen) must be ≤3 days prior to randomization
4. Subjects with adequate liver and renal function
5. Agree to the collection of nasopharyngeal swabs and venous blood
6. The participant or legally authorized representative signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol

Exclusion Criteria:

1. Have SpO2 ≤ 93% on room air at sea level or PaO2/FiO2 < 300, or a respiratory rate ≥30 per minute, or a heart rate ≥125 per minute
2. Has been admitted to a hospital prior to randomization, or is hospitalized (inpatient) at randomization, due to COVID-19 or requires treatment with supplemental oxygen
3. Have known allergies to any of the components used in the formulation of the study drug or placebo
4. Suspected or proven serious, active bacterial, fungal, viral, or other infection (besides COVID-19) requiring systemic therapy and that in the opinion of the investigator could constitute a risk to the subject or study assessments when taking study drug or placebo
5. Have any co-morbidity anticipated to require surgery within <7 days, or that is considered life threatening within 30 days
6. Have received treatment with the anti-androgen agents or 5-alpha reductase inhibitors within 3 months of the first dose
7. Prior, current, or planned future use of any of the following treatments at screening: COVID-19 convalescent plasma, mAbs against SARS-CoV-2, IVIG (any indication), where prior use is defined as the past 30 days or less than 5 half-lives of the investigational product (which is longer) from screening
8. Are investigator site personnel directly affiliated with this study
9. Have received an investigational intervention for SARS-CoV-2 prophylaxis within 30 days prior to randomization

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 380 (Actual)
Dates: Start 2021-08-04 (Actual); Primary Completion 2022-09-02 (Actual); Study Completion 2023-08-02 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects requiring oxygen by Day 28 | 28days

SECONDARY OUTCOMES:
Percentage of subjects who experience the events(such as hospitalization,Death etc.) by Day 28. (not applicable for subjects whose countries require mild to moderate COVID-19 patients to be hospitalised, such as COVID-19 patients in mainland China) | 28days

CONTACTS AND LOCATIONS:
Overall Officials: Cristhieni Rodrigues, Principal Investigator — Hospital Santa Paula
Locations (1):
- Hospital Santa Paula, São Paulo, São Paulo, Brazil